CLINICAL TRIAL: NCT03258866
Title: The Clinical Randomized Controlled Study of Different Dose Rituximab in the Treatment of Primary Immune Thrombocytopenia
Brief Title: The Study of Different Dose Rituximab in the Treatment of ITP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTX 4v1 in ITP
Record Dates: First submitted 2017-08-18; First posted 2017-08-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic; Immune Thrombocytopenia
Keywords: thrombocytopenia; Immune Thrombocytopenia; purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia; Purpura | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): In group A, Rituximab was given with a fixed dose of 100 mg administered as an intravenous infusion weekly (on day 1, 8, 15 and 22).
  Interventions: Drug: Rituximab
- group B (Experimental): In group B, Rituximab was given with a single dose of 375mg/m2
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — given with a fixed dose of 100 mg administered as an intravenous infusion weekly (on day 1, 8, 15 and 22)
  Other Names: Mabthera
  Arms: group A
Drug: Rituximab — given with a single dose of 375mg/m2
  Other Names: Mabthera
  Arms: group B

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University in China. In order to compare the efficacy, safety and response duration of different dose of rituximab in patients primary immune thrombocytopenia(pITP).

DETAILED DESCRIPTION:
62 patients with pITP who had failed to respond to glucocorticosteroids were randomly divided into 2 groups: group A(n = 32) and group B(n = 30). In group A, Rituximab was given with a fixed dose of 100 mg administered as an intravenous infusion weekly (on day 1, 8, 15 and 22). In group B, Rituximab was given with a single dose of 375mg/m2. The clinical effect, onset time, duration of efficacy and adverse reactions were observed to compare the efficacy and safety of two different plans.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for immune thrombocytopenia.
2. Male or female, between the ages of 10 ~ 70 years.
3. Normal glucocorticoid therapy is ineffective or effective but the maintenance dose is large, without immunosuppressive therapy or immunosuppressive treatment ineffective
4. To show a platelet count < 30×10^9/L, or with bleeding manifestations.
5. Eastern Cooperative Oncology Group（ECOG）performance status ≤ 2

Exclusion Criteria:

1. Current HIV infection or hepatitis B virus or hepatitis C virus infections.
2. Severe medical condition (lung, hepatic or renal disorder) other than ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)
3. Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period.
4. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.
5. Patients who are deemed unsuitable for the study by the investigator.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of platelet response(continuous response rate) | up to 1 year per subject
  Complete Response:a sustained (≥ 3 months) platelet count≥100×10^9/L;response: a sustained (≥ 3 months) platelet count ≥ 30×10^9/L without recurrence of thrombocytopenia;No response (NR): platelet count < 30 × 10^9/L or a less than two fold increase in platelet count from baseline or the presence of bleeding. Platelet count must be measured on two occasions more than a day apart.

SECONDARY OUTCOMES:
therapy associated adverse events | up to 1 year per subject
  The number and frequency of therapy associated adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, Dr, Principal Investigator — Shandong University
Locations (1):
- Qilu hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Auger S, Duny Y, Rossi JF, Quittet P. Rituximab before splenectomy in adults with primary idiopathic thrombocytopenic purpura: a meta-analysis. Br J Haematol. 2012 Aug;158(3):386-98. doi: 10.1111/j.1365-2141.2012.09169.x. Epub 2012 May 22. PMID 22612239
- [Background] Zaja F, Volpetti S, Chiozzotto M, Puglisi S, Isola M, Buttignol S, Fanin R. Long-term follow-up analysis after rituximab salvage therapy in adult patients with immune thrombocytopenia. Am J Hematol. 2012 Sep;87(9):886-9. doi: 10.1002/ajh.23272. Epub 2012 Jun 20. PMID 22718483
- [Result] Grace RF, Bennett CM, Ritchey AK, Jeng M, Thornburg CD, Lambert MP, Neier M, Recht M, Kumar M, Blanchette V, Klaassen RJ, Buchanan GR, Kurth MH, Nugent DJ, Thompson AA, Stine K, Kalish LA, Neufeld EJ. Response to steroids predicts response to rituximab in pediatric chronic immune thrombocytopenia. Pediatr Blood Cancer. 2012 Feb;58(2):221-5. doi: 10.1002/pbc.23130. Epub 2011 Jun 14. PMID 21674758
- [Result] Reboursiere E, Fouques H, Maigne G, Johnson H, Chantepie S, Gac AC, Reman O, Macro M, Benabed K, Troussard X, Damaj G, Cheze S. Rituximab salvage therapy in adults with immune thrombocytopenia: retrospective study on efficacy and safety profiles. Int J Hematol. 2016 Jul;104(1):85-91. doi: 10.1007/s12185-016-1992-4. Epub 2016 Apr 4. PMID 27040278
- [Result] Zaja F, Vianelli N, Volpetti S, Battista ML, Defina M, Palmieri S, Bocchia M, Medeot M, De Luca S, Ferrara F, Isola M, Baccarani M, Fanin R. Low-dose rituximab in adult patients with primary immune thrombocytopenia. Eur J Haematol. 2010 Oct;85(4):329-34. doi: 10.1111/j.1600-0609.2010.01486.x. Epub 2010 Jul 28. PMID 20546023
- [Result] Garcia-Suarez J, Prieto A, Reyes E, Manzano L, Merino JL, Alvarez-Mon M. The clinical outcome of autoimmune thrombocytopenic purpura patients is related to their T cell immunodeficiency. Br J Haematol. 1993 Jul;84(3):464-70. doi: 10.1111/j.1365-2141.1993.tb03102.x. PMID 8217798
- [Result] Gudbrandsdottir S, Birgens HS, Frederiksen H, Jensen BA, Jensen MK, Kjeldsen L, Klausen TW, Larsen H, Mourits-Andersen HT, Nielsen CH, Nielsen OJ, Plesner T, Pulczynski S, Rasmussen IH, Ronnov-Jessen D, Hasselbalch HC. Rituximab and dexamethasone vs dexamethasone monotherapy in newly diagnosed patients with primary immune thrombocytopenia. Blood. 2013 Mar 14;121(11):1976-81. doi: 10.1182/blood-2012-09-455691. Epub 2013 Jan 4. PMID 23293082
- [Result] Brah S, Chiche L, Fanciullino R, Bornet C, Mancini J, Schleinitz N, Jean R, Kaplanski G, Harle JR, Durand JM. Efficacy of rituximab in immune thrombocytopenic purpura: a retrospective survey. Ann Hematol. 2012 Feb;91(2):279-85. doi: 10.1007/s00277-011-1283-3. Epub 2011 Jun 28. PMID 21710166
- [Derived] Ni X, Li D, Yuan C, Yu Y, Wang H, Wang L, Yu T, Qin P, Peng J, Hou M, Shi Y, Hou Y. Single-dose versus low-dose rituximab in corticosteroid-resistant or relapsed ITP: A multicenter, randomized, controlled study. Am J Hematol. 2022 Apr;97(4):440-447. doi: 10.1002/ajh.26473. Epub 2022 Jan 25. PMID 35049070